CLINICAL TRIAL: NCT03194945
Title: Effects of Linagliptin and Metformin Monotherapy or Combined Sequential Treatment After Early Short-term Intensive Insulin Treatment on Long-term Blood Glucose Control and Function of β Cells in Patients With Type 2 Diabetes
Brief Title: Effects of Sequential Treatment Based on Lina/MET After Short-term Intensive Insulin in Newly Diagnosed Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Guangdong Provincial People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Dongguan People's Hospital (Other Government); Clifford Hospital (Unknown); Guangzhou Panyu Central Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Chinese PLA General Hospital (Other); Peking University People's Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai Changzheng Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Huizhou Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, Yanbing Li, Director of Endocrinology and Metabolism Department, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016146
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Continuous subcutaneous insulin infusion; Metformin; Linagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Linagliptin plus metformin (Active Comparator): CSII followed by Linagliptin 5 mg Qd + Metformin 0.5 g bid for 48 weeks
  Interventions: Drug: CSII followed by Lina+MET
- Linagliptin (Active Comparator): CSII followed by Linagliptin 5mg Qd for 48 weeks
  Interventions: Drug: CSII followed by Lina
- Metformin (Active Comparator): CSII followed by Metformin 0.5 bid for 48 weeks
  Interventions: Drug: CSII followed by MET
- Lifestyle alone (Active Comparator): No OHA is given after CSII
  Interventions: Drug: CSII alone

INTERVENTIONS:
Drug: CSII followed by Lina+MET — short-term intensive CSII followed by Linagliptin 5mg qd and Metformin 0.5g bid for 48 weeks
  Other Names: CSII+Lina+Met
  Arms: Linagliptin plus metformin
Drug: CSII followed by Lina — short-term intensive CSII followed by Linagliptin 5mg qd for 48 weeks
  Other Names: CSII+Lina
  Arms: Linagliptin
Drug: CSII followed by MET — short-term intensive CSII followed by Metformin 0.5g bid for 48 weeks
  Other Names: CSII+Met
  Arms: Metformin
Drug: CSII alone — No OHA is given after short-term intensive CSII
  Other Names: CSII
  Arms: Lifestyle alone

SUMMARY:
Short-term intensive insulin therapy(SIIT) is able to reverse β cell dysfunction and induce glycemic remission in patients with newly diagnosed type 2 diabetes. However, proportion of patients with response gradually decreases over time. There is no consensus on which treatment should be given in order to maintain the benefit in glycemic control and β cell recovery. In this multi-center, randomized, controlled study, effects of various sequential treatments ( metformin, linagliptin and combined with both drugs) on long-term blood glucose control as well as preservation of β cell function after SIIT were investigated.

In total, 412 patients with newly diagnosed type 2 diabetes who meet the inclusive criteria will be enrolled in eight centers in China. After baseline assessments, all patients will be treated with insulin pump to achieve and maintain euglycemia for 2 weeks. After completion of intensive treatment, insulin pump will be stopped. Different treatments will be applied to patients for 48 weeks according to randomization: Group A: Linagliptin 5 mg Qd + Metformin 0.5 g bid; Group B: Linagliptin 5 mg Qd; Group C: Metformin 0.5 g bid; Group D: No oral drugs. Primary endpoint is proportion of patients achieving glycosylated hemoglobin A1C <7% at the end of the study. Secondary endpoints include proportion of patients achieving glycosylated hemoglobin A1C <6.5% at the end of study; differences in β-cell function , insulin sensitivity, GLP-1 and glucagon secretion among treatment groups, and differences in adverse events among treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes who have never received any hypoglycemic treatment；
2. Fasting plasma glucose (FPG) between 7.0 mmol/l (126 mg/dl) and 16.7 mmol/l (300 mg/dl);
3. glycosylated hemoglobin A1C≥8.5%;
4. Aged between 20 and 70 years 5） body mass index (BMI) 22-35 kg/m2.

Exclusion Criteria:

1. Type 1 diabetes or special type of diabetes;
2. Acute complications of diabetes (including DKA, HHS and lactic acidosis)
3. Serious microvascular complications: proliferative stage of retinopathy; urine AER >300 mg/g or urine protein positive, quantification >0.5 g/d; uncontrolled painful diabetic neuropathy and significant diabetic autonomic neuropathy;
4. Severe macrovascular complications: acute cerebrovascular accident, acute coronary syndrome, vascular intervention for peripheral arterial disease or amputation requiring hospitalization within 12 months prior to enrollment;
5. Persistently increased blood pressure >180/110 mmHg;
6. Blood creatinine clearance less than 50 ml/min, alanine aminotransferase ≥2.5×upper limit of normal, total bilirubin ≥1.5×upper limit of normal;
7. Hemoglobin <100 g/L or need regular blood transfusion;
8. Use of drugs that may influence blood glucose within 12 weeks;
9. Systemic infection or serious concomitant disease; patients with malignancy or chronic diarrhea;
10. Uncontrolled endocrine gland dysfunction;
11. Patients with mental or communication disorders;
12. Chronic cardiac insufficiency, heart function class III and above;
13. Pregnant women, lactating women and women of child bearing age who are not willing to take contraception during the study;
14. Subjects who don't cooperate, cannot be followed up or have difficulty in completing the study considered by the investigator.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of subjects with optimal glycemic control | 48 weeks
  proportion of patients achieving glycosylated hemoglobin A1C <7% at the end of sequential treatment in each treatment group.

SECONDARY OUTCOMES:
proportion of subjects with excellent glycemic control | 48 weeks
  proportion of patients achieving glycosylated hemoglobin A1C <6.5% at the end of sequential treatment in each treatment group.
Change of β cell function | 48 weeks
  Differences in β-cell indicators among treatment arms at the end of study.
Change of insulin sensitivity | 48 weeks
  Differences in insulin sensitivity indicators among treatment arms at the end of study.
Incidence of adverse events | 48 weeks
  Differences in incidence of adverse events among treatment arms at the end of study.

CONTACTS AND LOCATIONS:
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu L, Ke W, Li H, Li F, Fan G, Kuang J, Ma J, Zhang X, Ji B, Li S, Du Y, Xue Y, Lyu Z, Gao L, Qu S, Shi Y, Yan L, Deng W, Xu C, Dai P, Xu L, Liu J, Wan X, Wei G, Yu S, Hong S, Zhang P, Huang Z, Cao X, Liao Z, Xiao H, Mu Y, Handelsman Y, Li Y. Intense simplified strategy for newly diagnosed type 2 diabetes in patients with severe hyperglycaemia: multicentre, open label, randomised trial. BMJ. 2024 Oct 15;387:e080122. doi: 10.1136/bmj-2024-080122. PMID 39406449